CLINICAL TRIAL: NCT01140997
Title: A Multi-center, Randomized, Open-label and Positive Controlled Phase II Clinical Trial to Assess Efficacy and Safety of Ypeginterferon Alfa-2b in Chronic Hepatitis C.
Brief Title: Efficacy and Safety of Ypeginterferon Alfa-2b in Chronic Hepatitis C
Acronym: PEGIFN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1006IFN
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; CHC; Hepatitis C, Chronic; Liver Diseases; Hepatitis, Chronic; Hepatitis, Viral, Human; Hepadnaviridae Infections; Antiviral Agents; Virus Diseases; Peginterferon alfa
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Diseases; Hepatitis, Chronic; Hepatitis, Viral, Human; Hepadnaviridae Infections; Virus Diseases | interventions — peginterferon alfa-2b; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Ypeginterferon alfa-2b 90mcg per Week, with Ribavirin 1000-1200mg/d
  Interventions: Drug: Ypeginterferon alfa-2b
- Group 2 (Experimental): Ypeginterferon alfa-2b 135mcg per Week, with Ribavirin 1000-1200mg/d
  Interventions: Drug: Ypeginterferon alfa-2b
- Group 3 (Experimental): Ypeginterferon alfa-2b 180mcg per Week, with Ribavirin 1000-1200mg/d
  Interventions: Drug: Ypeginterferon alfa-2b
- Group 4 (Active Comparator): Pegasys 180mcg per Week, with Ribavirin 1000-1200mg/d
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Ypeginterferon alfa-2b — sc, qw, for 48 weeks.
  Other Names: Peginterferon alfa-2b
  Arms: Group 1; Group 2; Group 3
Drug: Peginterferon alfa-2a — sc, qw, for 48 weeks.
  Other Names: Pegasys
  Arms: Group 4

SUMMARY:
This study is a multi-center, randomized, open-label and positive controlled Phase II Clinical trial to assess the efficacy and safety of Ypeginterferon alfa-2b (with Ribavirin), once a week, in 3 dose-groups respectively, for treatment of Chronic Hepatitis C patients, with Pegasys 180mcg/week & Ribavirin as positive control. It is aimed to establish a dose response and safety relationship sufficient to allow the subsequent design and conduct of Phase III trials, and generate the PK data in hepatitis C patients to satisfy regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~65 years.
* Pregnancy tests of female patients must be negative. All patients with effective birth control measures during treatment period and 6 months after the cessation of treatment.
* Chronic HCV infection evidence: HCV RNA or anti-HCV positive >6 months; liver biopsy evidence; vital signs, symptoms, exposure history, and results of laboratory test and iconography examination support diagnosis of chronic hepatitis C.
* HCV RNA≥2000IU/ml.

Exclusion Criteria:

* Pregnant or lactating women.
* Mental disorder or physical disability.
* WBC<3000/mm3, or ANC <1500/mm3, or PLT <90,000/mm3.
* Received interferon treatment within the previous 6 months or shew no response to interferon.
* Co-infection with HIV, HAV, HBV, HEV.
* Evidence of hepatic decompensation.
* Chest X-ray with clinically significant active inflammatory process, history of significant pulmonary disease or any history of interstitial lung disease.
* History of hypothyroidism or current treatment for thyroid disease.
* Diabetes mellitus.
* Uncontrolled significant chronic medical conditions other than chronic hepatitis C or other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | week 12
  Proportion of patients with HCV RNA undetectable at week 12.

SECONDARY OUTCOMES:
Efficacy | Week 4, 12, 24, 48 and 72
  1. Proportion of patients with HCV RNA undetectable at Week 4, 24,48 and 72;
  2. Average decline level of log10 of HCV RNA at Week 4, 12, 24, 48 and 72.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lai, MD, PhD, Principal Investigator — Peking University People's Hospital
Locations (38):
- China (38):
  - 302 Military Hospital, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Youyi Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - First Affiliated Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central-south University, Changsha
  - Xiangya Second Hospital, Central-south University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Southwest Hospital, Chongqing
  - Fuzhou Infectious Disease Hospital, Fuzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - Nangfang Hospital, Guangzhou
  - First Affiliated Hospital of Guangxi Medical Universtiy, Guilin
  - Second Affiliated Hospital of Harbin Medical University, Harbin
  - First Affiliated Hospital of Anhui Medical University, Hefei
  - Jinan Infectious Disease Hospital, Jinan
  - First Affiliated Hospital of Lanzhou University, Lanzhou
  - First Affiliated Hospital of Nanchang University, Nanchang
  - 81 Military Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Second Hospital of Nanjing, Nanjing
  - 85 Military Hospital, Shanghai
  - Changhai Hospital, Shanghai
  - Huashan Hospital, Shanghai
  - Renji Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Shenzhen Third People's Hospital, Shenzhen
  - Third Affiliated Hospital, Hebei Medical University, Shijiazhuang
  - First Affiliated Hospital, Shanxi University, Taiyuan
  - Tianjin Third Central Hospital, Tianjin
  - First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - Tongji Hospital, Huazhong University of Science&Technology, Wuhan
  - Tangdu Hospital, Fouth Military Medical University, Xi'an
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou

REFERENCES:
- [Derived] Feng B, Yang RF, Xie Q, Shang J, Kong FY, Zhang HY, Rao HY, Jin Q, Cong X, Liu YY, Kang Y, Wei L. Hepatitis C virus core antigen, an earlier and stronger predictor on sustained virological response in patients with genotype 1 HCV infection. BMC Gastroenterol. 2014 Mar 13;14:47. doi: 10.1186/1471-230X-14-47. PMID 24625322